CLINICAL TRIAL: NCT03286673
Title: Comparison of Three Calcium Supplements With Regard to Their Metabolic Effects in Healthy Adults
Brief Title: Comparison of Three Calcium Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. Gerhard Jahreis, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H28-06
Record Dates: First submitted 2017-09-11; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: calcium carbonate; calcium phosphate; metabolic effects; human study; calcium and phosphorus metabolism
MeSH Terms: interventions — calcium phosphate; tricalcium phosphate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- calcium phosphate (Experimental): Pentacalcium hydroxy-triphosphate (Ca5(PO4)3OH) was incorporated in wholemeal and crispy wafer bread in order to achieve a additional calcium intake of 1000 mg/d.
  Interventions: Dietary Supplement: calcium phosphate
- Tricalcium Phosphate (Experimental): β-tricalcium phosphate (Ca3(PO4)2) as incorporated in wholemeal and crispy wafer bread in order to achieve a additional calcium intake of 1000 mg/d.
  Interventions: Dietary Supplement: Tricalcium Phosphate
- Calcium carbonate (Experimental): Calcium carbonate (CaCO3) was incorporated in wholemeal and crispy wafer bread in order to achieve a additional calcium intake of 1000 mg/d.
  Interventions: Dietary Supplement: Calcium carbonate
- Placebo (Active Comparator): Wholemeal and crispy wafer bread without additional calcium additive.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: calcium phosphate
  Arms: calcium phosphate
Dietary Supplement: Tricalcium Phosphate
  Arms: Tricalcium Phosphate
Dietary Supplement: Calcium carbonate
  Arms: Calcium carbonate
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The study was conducted to investigate the metabolic effects of three different calcium compounds in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 40 years

Exclusion Criteria:

* diseases of the gastrointestinal tract
* pregnancy
* the intake of any medication (e. g. for thyroid gland)
* intake of dietary supplements

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Serum mineral concentration | after 4 weeks of each intervention
  Calcium and Phosphate (and others) concentration in serum.
Stool mineral concentration | after 4 weeks of each intervention
  Calcium and Phosphate concentration (and others) in stool from a three day stool collection
Urine mineral concentration | after 4 weeks of each intervention
  Calcium and Phosphate concentration (and others) in urine from a three day urine collection
Lipids in blood | after 4 weeks of each intervention
  Lipids and lipoprotein concentration in serum.
Sterols | after 4 weeks of each intervention
  Neutrals sterols and bile acids in stool from a three day stool collection
Dietary intake | after 4 weeks of each intervention
  Evaluation of the dietary intake using a three day weighed dietary record.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition

IPD SHARING:
Plan to Share IPD: No